CLINICAL TRIAL: NCT05913596
Title: A Multicenter, Prospective, One-arm Clinical Study
Brief Title: The Safety and Efficacy of CD38 Monoclonal Antibody Monotherapy for CaAMR in Renal Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20220103C-R1
Record Dates: First submitted 2023-03-29; First posted 2023-06-22 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-03

CONDITIONS: Antibody-mediated Rejection; Kidney Tranplant
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Each patient received CD38 monoclonal antibody monotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with CaAMR (Experimental): This is a multicenter, prospective, single arm clinical study. The study will enroll 15 renal transplant recipients with positive DSA and CaAMR confirmed by biopsy after renal transplantation. According to inclusion and exclusion criteria patients will be screened to participate in the trial.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — After successful enrollment, the patient will receive daratumumab of 16mg/kg once every two weeks (0-22 weeks) for a total of 12 times. Peripheral blood samples were collected from 0 to 24 weeks (weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24) for routine blood tests, liver and kidney function electrolytes, tacrolimus or cyclosporine trough concentrations, HLA antibody quantification (weeks 0, 4, 8, 12, 16, 20, and 24), infection indicators (weeks 0, 8, and 24), immune status assessments (weeks 0, 4, 8, 12, 16, 20, and 24), and biopsy of transplanted kidneys was performed at 24 weeks to assess pathological changes.
  Other Names: CD38 monoclonal antibody

SUMMARY:
Renal transplantation is the best choice for the treatment of end-stage renal disease, but the long-term survival of the graft is still remains a challenge. Chronic antibody-mediated rejection (AMR) is the main factor affecting the long-term survival of the graft. There is still no effective treatment for chronic antibody-mediated rejection, even in the active phase (CaAMR). In recent years, new therapeutic drugs based on the generation of DSA and the mechanism of AMR, including protease inhibitor bortezomi, CD20 monoclonal antibody, C5 monoclonal antibody and IL-6 antibody, have not been able to effectively eliminate and inhibit the generation of DSA, nor have they been proved to have a definite effect on AMR.

CD38 is a type II transmembrane protein that is highly expressed on plasma cells and NK cells, which are considered to play a key role in the occurrence and development of AMR. Recently, a few cases have reported that CD38 monoclonal antibody combined plasma exchange and/or IVIG may be an effective strategy for the prevention and treatment of AMR, but the effectiveness and safety of daratumumab monotherapy on CaAMR were unknown. This is a multicenter, prospective, single arm clinical study. The study will enroll 15 renal transplant recipients with positive DSA and CaAMR confirmed by biopsy after renal transplantation. According to inclusion and exclusion criteria patients will be screened to participate in the trial.

DETAILED DESCRIPTION:
After successful enrollment, the patient will receive daratumumab of 16mg/kg once every two weeks (0-22 weeks) for a total of 12 times, and continue to receive triple immunosuppressive therapy with prednisone, mycophenolic acid, tacrolimus (target valley concentration of 5-7ng/ml) or cyclosporine (target valley concentration of 100-200ng/ml). Peripheral blood samples were collected from 0 to 24 weeks (weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24) for routine blood tests, liver and kidney function electrolytes, tacrolimus or cyclosporine trough concentrations, HLA antibody quantification (weeks 0, 4, 8, 12, 16, 20, and 24), infection indicators (weeks 0, 8, and 24), immune status assessments (weeks 0, 4, 8, 12, 16, 20, and 24), and biopsy of transplanted kidneys was performed at 24 weeks to assess pathological changes.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of written informed consent
2. Age ≥ 18 years old
3. ≥ 180 days after living donor kidney or DD donor kidney transplantation
4. EGFR ≥ 30mL/min/1.73 m2 (CKD-EPI formula)
5. Pre stored and/or newborn DSA (HLA antibody)

Exclusion Criteria:

1. Patients participating in another clinical trial
2. Age less than 18 years old
3. Female subjects are pregnant or breastfeeding, or do not receive appropriate contraceptive measures
4. ABO incompatibility transplantation
5. Kidney transplantation biopsy combined with one of the following results:

   A. T-cell mediated rejection B. New or recurrent severe thrombotic microangiopathy C. Polyomavirus nephropathy
6. Receive anti acute rejection treatment within 3 months before screening
7. Have been treated with other immunomodulatory monoclonal/polyclonal antibodies (such as CD20 antibody, bortezomib, C5 monoclonal antibody, IL-6/IL-6R antibody) within 3 months
8. Total bilirubin>2 times the upper normal limit, alanine aminotransferase and aspartate aminotransferase>2.5 times the upper normal limit
9. Hemoglobin<8 g/dL
10. Thrombocytopenia: Platelets<100 × 109/L
11. Leukopenia: White blood cells<3 × 109/L, neutropenia: neutrophils<1.5 × 109/L
12. Hypogammaglobulinemia: Serum IgG<400 mg/dL
13. Eliminate active viral, bacterial, or fungal infections
14. Excluding Active Malignant Diseases with Intensive Immunosuppressive Therapy
15. Latent or active tuberculosis
16. Inoculate live vaccine within 6 weeks after screening
17. History of alcohol or illicit drug abuse
18. Serious medical or mental illness that may affect participation in the study
19. Active hepatitis B virus infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
The change of donor specific antibody | 6 months
  Donor specific antibody changed 30% based on luminex HLA testing

SECONDARY OUTCOMES:
The change of serum creatinine | 6 months
  Creatinine changed by 30% compared to before treatment or returned to baseline level
The change of BANFF score | 6 months
  The change of BANFF score, including c, g, ptc score
Incidence of treatment-related adverse events | 6 months
  Adverse event monitoring, assessment of labs, monitoring of viral PCRs
The change of NK cell count in PBMC | 6 months
  The change of NK cell count in PBMC collected at multiple time points throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Wu, MD, Principal Investigator — the First Affiliated Hospital of Medicine College, Zhejiang University
Locations (1):
- 79# Qingchun Road, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators will disclose our research protocol, the clinical outcome of the investigator, and the original data of the participants can be obtained by contacting the investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the end of the study
Access Criteria: Contact the investigator to obtain via email